CLINICAL TRIAL: NCT04793620
Title: A Phase 1, Randomized, Double Blind, Active-Controlled Dose-Escalation Study to Assess the Safety and Immunogenicity of Pertussis Acellular Vaccine Adjuvanted With TQL1055 (PAVA)
Brief Title: Pertussis Acellular Vaccine Adjuvanted With TQL1055
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: financial constraints
Sponsor: Adjuvance Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: V1.1-101
Record Dates: First submitted 2021-03-04; First posted 2021-03-11 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Pertussis
Keywords: vaccine; adjuvant
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Intervention Model Description: Sequential-group dose-escalation study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQL1055 (Experimental): TQL1055 + acellular pertussis vaccine
  Interventions: Other: TQL1055; Biological: Acellular pertussis vaccine
- Acellular pertussis vaccine (Active Comparator): Acellular pertussis vaccine
  Interventions: Biological: Acellular pertussis vaccine

INTERVENTIONS:
Other: TQL1055 — Semisynthetic saponin adjuvant
  Arms: TQL1055
Biological: Acellular pertussis vaccine — Acellular pertussis vaccine

SUMMARY:
This is a phase 1 study to evaluate the safety and immunogenicity of the semisynthetic saponin adjuvant TQL1055 administered in combination with an acellular pertussis vaccine.

DETAILED DESCRIPTION:
The recent increase in the incidence of pertussis has prompted the need for improvements to current acellular pertussis vaccines. Use of novel adjuvants is one approach to such improvement. TQL1055 is a rationally designed, semisynthetic analog of the licensed Quillaja saponin (QS)-21. It has been designed to maintain adjuvant activity with improved tolerability and greater ease of manufacture.

This is a Phase 1, randomized, double blind, active-controlled sequential-group study, designed to evaluate the safety, tolerability, and immunogenicity of the combination of TQL1055 and acellular pertussis vaccine. The dose of TQL1055 will increase by group.

ELIGIBILITY:
Key Inclusion Criteria:

* 18 to 50 years of age
* General good health
* BMI between 17 and 35 kg/m2
* Not of childbearing potential OR using adequate contraception

Key Exclusion Criteria:

* Pregnant or lactating
* Prior medical condition that could adversely affect subject safety
* Clinically significant abnormal laboratory parameter
* Current acute febrile illness
* Contraindication to intramuscular injection
* Contraindication to pertussis vaccination
* Received pertussis vaccine within 3 years

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Reactogenicity | 7 days
  Solicited local and systemic adverse events

SECONDARY OUTCOMES:
Adverse Events | 365 days
  Adverse Events/Serious Adverse Events
Incidence of abnormal laboratory test results | 28 days
  Incidence of abnormal laboratory test results
Immunogenicity | 28 days
  Anti-Pertussis Toxin antibodies
Immunogenicity | 365 days
  Anti-Pertussis Toxin antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Sean R Bennett, MD PhD, Study Director — Adjuvance Technologies, Inc.
Locations (1):
- Q-Pharm, Brisbane, Australia

IPD SHARING:
Plan to Share IPD: No